CLINICAL TRIAL: NCT01822496
Title: A Randomized Phase II Study of Individualized Combined Modality Therapy for Stage III Non-small Cell Lung Cancer (NSCLC)
Brief Title: Erlotinib Hydrochloride or Crizotinib and Chemoradiation Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00737; NCI-2013-00737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-1306 (Other: NRG Oncology); RTOG-1306 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2013-04-01; First posted 2013-04-02 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Stage III Non-Small Cell Lung Cancer AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Crizotinib; Erlotinib Hydrochloride; Etoposide; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EGFR: Erlotinib (Experimental): Induction erlotinib for 12 weeks followed by chemotherapy (either cisplatin/etoposide or paclitaxel/carboplatin) and radiation therapy. Patients who have had no response (partial or complete) after 6 weeks of induction therapy start chemoradiation therapy immediately.
  Interventions: Radiation: Radiation Therapy; Drug: Carboplatin; Drug: Cisplatin; Drug: Erlotinib; Drug: Etoposide; Drug: Paclitaxel
- EGFR: No Erlotinib (Active Comparator): Chemotherapy (either cisplatin/etoposide or paclitaxel/carboplatin) and radiation therapy.
  Interventions: Radiation: Radiation Therapy; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Paclitaxel
- ALK: Crizotinib (Experimental): Induction crizotinib for 12 weeks followed by chemotherapy (either cisplatin/etoposide or paclitaxel/carboplatin) and radiation therapy. Patients who have had no response (partial or complete) after 6 weeks of induction therapy start chemoradiation therapy immediately.
  Interventions: Radiation: Radiation Therapy; Drug: Carboplatin; Drug: Cisplatin; Drug: Crizotinib; Drug: Etoposide; Drug: Paclitaxel
- ALK: No Crizotinib (Active Comparator): Chemotherapy (either cisplatin/etoposide or paclitaxel/carboplatin) and radiation therapy.
  Interventions: Radiation: Radiation Therapy; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Radiation Therapy — 30 once-daily 2 Gy fractions over 6 weeks totaling 60 Gy of intensity-modulated radiation therapy (IMRT) or 3-dimensional conformal radiation therapy (3D-CRT).
  Other Names: 3-dimensional conformal radiation therapy; 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; IMRT; Intensity-modulated radiation therapy
Drug: Carboplatin — Concurrent: AUC=2, IV, days 1, 8, 14, 22, 29, and 36 of radiation therapy. For patients receiving either erlotinib or crizotinib, carboplatin will begin 2 weeks after erlotinib or crizotinib, as applicable.
  Consolidation: 4-6 weeks after completion of RT, AUC=6, IV, days 1 and 22.
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — 50 mg/m2, IV (intravenous), on days 1 and 8 of two 4-week cycles concurrent with radiation therapy. For patients receiving either erlotinib or crizotinib, cisplatin will begin 2 weeks after the completion of erlotinib or crizotinib, as applicable.
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Crizotinib — 250 mg, orally, twice daily for four 3-week cycles (12 weeks in total)
  Other Names: MET Tyrosine Kinase Inhibitor PF-02341066; PF-02341066; PF-2341066; Xalkori
  Arms: ALK: Crizotinib
Drug: Erlotinib — 150 mg, orally, once daily for four 3-week cycles (12 weeks in total)
  Other Names: Cp-358,774; Erlotinib Hydrochloride; OSI-774; Tarceva
  Arms: EGFR: Erlotinib
Drug: Etoposide — 50 mg/m2, IV, on days 1 and 8 of two 4-week cycles concurrent with radiation therapy. For patients receiving either erlotinib or crizotinib, etoposide will begin 2 weeks after the completion of erlotinib or crizotinib, as applicable.
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Paclitaxel — Concurrent: 45 mg/m2, IV, days 1, 8, 14, 22, 29, and 36 of radiation therapy. For patients receiving either erlotinib or crizotinib, carboplatin will begin 2 weeks after erlotinib or crizotinib, as applicable.
  Consolidation: 4-6 weeks after completion of RT, 200 mg/m2, IV, days 1 and 22.
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This randomized phase II trial studies how well erlotinib hydrochloride or crizotinib with chemoradiation therapy works in treating patients with stage III non-small cell lung cancer. Radiation therapy uses high energy x rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin, etoposide, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving erlotinib hydrochloride is more effective than crizotinib with chemoradiation therapy in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether patients with unresectable local-regionally advanced non-small cell lung cancer (NSCLC) treated with targeted agents based on molecular characteristics have a longer progression-free survival than those treated with standard care therapy alone.

SECONDARY OBJECTIVES:

I. To evaluate response rate. II. To assess toxicity. III. To assess overall survival. IV. To correlate clinical outcomes with tumor molecular aberrations identified from deep sequencing of selected kinomes in patients from whom adequate baseline tissue is available.

OUTLINE: Eligible patients are assigned to one of two cohorts based on pre-enrollment screening by the enrolling institution for two biomarkers: EGFR TK mutation and EML4-ALK fusion arrangement. Within each cohort, patients are randomized to either an experimental or control arm, resulting in a total of four treatment arms overall. Patients with both the EGFR mutation and ALK arrangement are placed in the ALK Cohort.

Planned Sample Size: 156 for the EGFR mutation cohort and 78 for the ALK translocation cohort

After completion of study treatment, patients are followed at 1 and 2 months, 4-6 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, newly diagnosed non-squamous NSCLC
* Unresectable stage IIIA or IIIB disease; patients must be surgically staged to confirm N2 or N3 disease; patients may have invasive mediastinal staging by mediastinoscopy, mediastinotomy, endobronchial ultrasound transbronchial aspiration (EBUS-TBNA), endoscopic ultrasound (EUS), or video-assisted thoracoscopic surgery (VATS)
* Patients with any tumor (T) with node (N)2 or N3 are eligible; patients with T3, N1-N3 disease are eligible if deemed unresectable; patients with T4, any N are eligible
* Patients must have measurable disease, i.e., lesions that can be accurately measured in at least 1 dimension (longest dimension in the plane of measurement is to be recorded) with a minimum size of 10 mm by computed tomography (CT) scan (CT scan slice thickness no greater than 5 mm)
* Patients with a pleural effusion, which is a transudate, cytologically negative and non-bloody, are eligible if the radiation oncologist feels the tumor can be encompassed within a reasonable field of radiotherapy
* If a pleural effusion can be seen on the chest CT but not on chest x-ray and is too small to tap, the patient will be eligible; patients who develop a new pleural effusion after thoracotomy or other invasive thoracic procedure will be eligible
* The institution's pre-enrollment biomarker screening at a Clinical Laboratory Improvement Amendments (CLIA) certified lab documents presence of known "sensitive" mutations in epidermal growth factor receptor tyrosine kinase (EGFR TK) domain (exon 19 deletion, L858) and/or EML4-anaplastic lymphoma kinase (ALK) fusion arrangement; either the primary tumor or the metastatic lymph node tissue may be used for testing of mutations
* The institution's pre-enrollment biomarker screening at a CLIA certified lab documents absence of T790M mutation in the EGFR TK domain
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination, including recording of pulse, blood pressure (BP), weight, and body surface area, within 45 days prior to registration
  * Whole body fludeoxyglucose-positron emission tomography (FDG-PET)/CT (orbits to mid-thighs) within 30 days prior to registration; PET/CT must be negative for distant metastasis
  * CT scan with contrast of the chest and upper abdomen to include liver and adrenals (unless medically contraindicated) within 30 days prior to registration
  * Magnetic resonance imaging (MRI) of the brain with contrast (or CT scan with contrast, if MRI medically contraindicated) within 30 days prior to registration
* Zubrod performance status 0-1 within 14 days prior to registration
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 8.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Serum creatinine < 1.5 mg/dL or calculated creatinine clearance >= 50 ml/min (by Cockcroft-Gault formula) within 14 days prior to registration
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) within 14 days prior to registration
* Bilirubin within normal institutional limits within 14 days prior to registration
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* Patient must provide study specific informed consent prior to study entry, including consent for mandatory screening of tissue

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 730 days (2 years) (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Atelectasis of the entire lung
* Contralateral hilar node involvement
* Exudative, bloody, or cytologically malignant effusions
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; protocol-specific requirements may also exclude immuno-compromised patients
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Prior allergic reaction to the study drug(s) involved in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, Principal Investigator — NRG Oncology
Locations (174):
- United States (174):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - AMITA Health Cancer Institute and Outpatient Center, Hinsdale, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Concord Hospital, Concord, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Intermountain Medical Center, Murray, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Started | 16 | 23 | 9 | 11
Eligible | 14 | 21 | 9 | 7
Eligible With Disease Assessment | 10 | 15 | 6 | 4
Eligible and Started Study Treatment | 14 | 20 | 9 | 7
Completed (Subjects contributing any data to results are considered to have completed the study) | 14 | 21 | 9 | 7
Not Completed | 2 | 2 | 0 | 4
Not completed — Protocol Violation | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib | Total
Number analyzed (Participants) | 14 | 21 | 9 | 7 | 51
Age, Customized [Count of Participants; unit: Participants]
  Age (years): ≤ 49 | 2 | 3 | 3 | 0 | 8
  Age (years): 50 - 59 | 4 | 5 | 4 | 2 | 15
  Age (years): 60 -69 | 4 | 9 | 2 | 1 | 16
  Age (years): ≥ 70 | 4 | 4 | 0 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 5 | 19
  Male | 10 | 15 | 5 | 2 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 13 | 19 | 9 | 6 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 12 | 15 | 7 | 5 | 39
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST) guideline v1.1 as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions at any location. Progression-free survival time is measured from the date of randomization to the date of first progression, death, or last known follow-up (censored). No statistical testing was done due to early study termination.
Time Frame: From randomization to study termination. Maximum follow-up was 39.0 months
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 14 | 21 | 9 | 7
months | 21.1 [8.5 to NA] — Not reached | 9.2 [8.7 to NA] — Not reached | 14.7 [6.4 to 19.5] | NA [NA to NA] — Not reached

2. Secondary Outcome: Percentage of Patients With Complete or Partial Response
Description: Per the RECIST guideline v1.1 complete response is defined as the disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. No statistical testing was done due to early study termination.
Time Frame: From randomization to study termination. Maximum follow-up was 39.0 months
Population: Eligible patients with disease assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 10 | 15 | 6 | 4
percentage of participants | 50.0 [19.0 to 81.0] | 26.7 [4.3 to 49.1] | 66.7 [29.0 to 100.0] | 75.0 [32.6 to 100.0]

3. Secondary Outcome: Number of Patients With Grade 3-5 Adverse Events
Description: Adverse events (AE) are graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From randomization to study termination. Maximum follow-up was 39.0 months
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 14 | 20 | 9 | 7
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From randomization to study termination. Maximum follow-up was 39.0 months
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 14 | 21 | 9 | 7
Months | NA [NA to NA] — Not reached | 35.9 [35.9 to NA] — Not reached | NA [NA to NA] — Not reached | NA [NA to NA] — Not reached

5. Secondary Outcome: Local-regional Progression-free Survival
Description: Progression is defined using the RECIST guideline v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new regional lesions. Local progression is defined as progression within the planning target volume (PTV). Regional progression is defined as progression outside of the PTV but within the same lobe of the lung as the primary tumor or in regional lymph nodes as defined by the American Joint Committee on Cancer (AJCC) 7th edition nodal stations. Local-regional progression-free survival time is measured from the date of randomization to the date of first local-regional progression, death, or last known follow-up (censored). Local-regional progression-free survival rates are estimated using the Kaplan-Meier method. No testing was done due to early study termination.
Time Frame: From randomization to study termination. Maximum follow-up was 39.0 months
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 14 | 21 | 9 | 7
Months | 25.7 [8.5 to NA] — Not reached | NA [NA to NA] — Not reached | 14.7 [6.4 to 19.5] | NA [NA to NA] — Not reached

6. Secondary Outcome: Distant Progression-free Survival
Description: Distant progression is defined as the first occurrence of distant metastasis. Distant progression-free survival time is measured from the date of randomization to the date of first distant progression, death, or last known follow-up (censored). Distant progression-free survival rates are estimated using the Kaplan-Meier method. No testing was done due to early study termination.
Time Frame: From randomization to study termination. Maximum follow-up was 39.0 months
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 14 | 21 | 9 | 7
Months | NA [NA to NA] — Not reached | 35.9 [8.9 to 35.9] | NA [NA to NA] — Not reached | 20.1 [7.8 to NA] — Not reached

7. Secondary Outcome: Correlation Between Clinical Outcomes and Tumor Molecular Aberrations
Time Frame: Baseline
Population: The data required for this analysis was not obtained and will not be obtained.
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Maximum follow-up was 39.0 months.
Description: Eligible patients who started treatment are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | EGFR: Erlotinib | EGFR: No Erlotinib | ALK: Crizotinib | ALK: No Crizotinib
All-Cause Mortality (participants affected / at risk) | 1/14 | 3/20 | 2/9 | 1/7
Serious Adverse Events (participants affected / at risk) | 1/14 | 7/20 | 4/9 | 2/7
Other Adverse Events (participants affected / at risk) | 14/14 | 20/20 | 8/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGFR: Erlotinib (N=14) | EGFR: No Erlotinib (N=20) | ALK: Crizotinib (N=9) | ALK: No Crizotinib (N=7)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Esophageal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Fever (General disorders) | 0 | 1 | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EGFR: Erlotinib (N=14) | EGFR: No Erlotinib (N=20) | ALK: Crizotinib (N=9) | ALK: No Crizotinib (N=7)
Anemia (Blood and lymphatic system disorders) | 8 | 10 | 4 | 6
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Endocrine disorders - Other (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Blurred vision (Eye disorders) | 2 | 2 | 2 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0
Eye disorders - Other (Eye disorders) | 2 | 0 | 0 | 0
Flashing lights (Eye disorders) | 0 | 0 | 0 | 1
Floaters (Eye disorders) | 1 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 8 | 1 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 11 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 8 | 10 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 5 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 8 | 6 | 1 | 4
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Esophageal stenosis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 10 | 12 | 4 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 0 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 16 | 6 | 4
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6 | 3 | 2
Chills (General disorders) | 1 | 2 | 0 | 0
Death NOS (General disorders) | 0 | 1 | 0 | 0
Edema face (General disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 2 | 1 | 4
Fatigue (General disorders) | 13 | 14 | 6 | 7
Fever (General disorders) | 5 | 1 | 1 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other (General disorders) | 1 | 2 | 0 | 1
Irritability (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 3 | 0 | 2
Pain (General disorders) | 3 | 1 | 0 | 3
Allergic reaction (Immune system disorders) | 1 | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 2 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 2 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Uterine infection (Infections and infestations) | 1 | 0 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 8 | 6 | 1 | 4
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 2 | 1
Alkaline phosphatase increased (Investigations) | 2 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 2 | 1
Blood bilirubin increased (Investigations) | 3 | 1 | 0 | 1
Creatinine increased (Investigations) | 2 | 5 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0
Investigations - Other (Investigations) | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 8 | 10 | 2 | 4
Neutrophil count decreased (Investigations) | 4 | 7 | 3 | 3
Platelet count decreased (Investigations) | 5 | 9 | 2 | 5
Weight gain (Investigations) | 1 | 1 | 0 | 1
Weight loss (Investigations) | 5 | 3 | 0 | 1
White blood cell decreased (Investigations) | 5 | 6 | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 6 | 9 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 4 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 6 | 2 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 2
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 5 | 3 | 3
Dysgeusia (Nervous system disorders) | 3 | 1 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 6 | 4 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 2 | 0 | 0 | 0
Olfactory nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 9 | 2 | 4
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 3 | 2 | 2
Depression (Psychiatric disorders) | 3 | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 4 | 3 | 2
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 2 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 3 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 12 | 4 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7 | 3 | 4
Body odor (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 3 | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 | 3 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 1 | 2 | 1 | 0
Hypertension (Vascular disorders) | 1 | 4 | 1 | 2
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0
Superficial thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 2 | 0 | 2

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 59 subjects accrued out of 234 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT01822496/Prot_SAP_000.pdf